CLINICAL TRIAL: NCT03107182
Title: A Phase II Trial of Nivolumab/Nab-paclitaxel/Carboplatin Induction Chemotherapy Followed by Response-stratified Locoregional Therapy for Patients With Locoregionally Advanced HPV-related Oropharyngeal Cancer- the OPTIMA II Trial
Brief Title: Chemotherapy and Locoregional Therapy Trial (Surgery or Radiation) for Patients With Head and Neck Cancer
Acronym: OPTIMA-II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-0104
Record Dates: First submitted 2017-03-29; First posted 2017-04-11 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: HPV-Related Squamous Cell Carcinoma; HNSCC
Keywords: HPV- positive HNSCC; head and neck squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — 130-nm albumin-bound paclitaxel; Taxes; Albumin-Bound Paclitaxel; Carboplatin; Nivolumab; Cisplatin; Hydroxyurea; Fluorouracil; Dexamethasone; Famotidine; Diphenhydramine; Paclitaxel; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Induction Chemotherapy (Experimental): All enrolled patients will receive three 21-day cycles of chemotherapy consisting of nab-paclitaxel (100 mg/m2 on days 1, 8, 15; 9 doses total), carboplatin (AUC 5 on day 1; 3 doses total), and nivolumab (360 mg on days 1; 3 doses total). Growth factor support will be provided using G-CSF administered on days 16-18.
  Adjuvant nivolumab will be offered to all patients for 6-months post completion of locoregional therapy.
  Interventions: Drug: nab-paclitaxel; Drug: Carboplatin; Drug: Nivolumab
- Single Modality De-escalation Arm (SDA) (Experimental): Following the induction treatments (carboplatin, nab-paclitaxel, and nivolumab), patients will be assessed based on response to chemotherapy and high or low risk status.
  Patients with low risk and small volume tonsillar disease (T1-T2, non-bulky N2A-N2B with ≤2 non-lower neck lymph nodes measuring ≤5 cm in size) or base of tongue disease (T1-2 with lateralized primary ≤3 cm, non-bulky N2A-N2B with ≤2 non-lower neck lymph nodes measuring ≤5 cm in size) who have ≥50% reduction by RECIST following induction chemotherapy will undergo TORS and selective nodal dissection. De-intensified adjuvant RT will be given for adverse pathologic features. Patients may refuse TORS treatment.
  Patients with low risk, who do not qualify for TORS (due to volume of disease or poor visualization/access) or refuse TORS, who have ≥50% reduction by RECIST following induction chemotherapy will be given de-intensified treatment with radiation alone to 50 G.
  Interventions: Drug: Nivolumab; Procedure: Transoral robotic surgery (TORS); Radiation: Adjuvant RT
- Intermediate De-escalation Arm (IDA) (Experimental): Following the induction treatments (carboplatin, nab-paclitaxel, and nivolumab), patients will be assessed based on response to chemotherapy and high or low risk status.
  Patients who have low risk disease with <50% but ≥30% reduction of tumor by RECIST with induction chemotherapy will receive CRT to 50 Gy with concurrent bolus cisplatin (x2 doses) or TFHX (paclitaxel, 5-FU, hydroxyurea, dexamethasone, famotidine, and diphenhydramine) to 45 Gy (3 cycles).
  Patients who have high risk disease and ≥50% reduction of tumor by RECIST with induction chemotherapy will receive CRT to 50 Gy with concurrent bolus cisplatin (x2 doses) or TFHX to 45 Gy (3 cycles).
  Interventions: Drug: Nivolumab; Drug: Cisplatin; Drug: Hydroxyurea; Drug: 5-FU; Drug: Dexamethasone; Drug: Famotidine; Drug: Diphenhydramine; Drug: Paclitaxel; Radiation: Chemoradiotherapy
- Regular Dose Arm (RDA) (Experimental): Following the induction treatments (carboplatin, nab-paclitaxel, and nivolumab), patients will be assessed based on response to chemotherapy and high or low risk status.
  Patients who have low risk disease and <30% reduction of tumor by RECIST with induction chemotherapy will receive CRT to 70 Gy with concurrent bolus cisplatin (x3 doses) or TFHX (paclitaxel, 5-FU, hydroxyurea, dexamethasone, famotidine, and diphenhydramine) to 75 Gy (5 cycles).
  Patients who have high risk disease and <50% reduction of tumor by RECIST with induction chemotherapy will receive CRT to 70 Gy with concurrent bolus cisplatin (x3 doses) or TFHX to 75 Gy (5 cycles).
  Any patient who has progressive disease will receive CRT to 70 Gy with concurrent bolus cisplatin (x3 doses) or TFHX to 75 Gy (5 cycles).
  Interventions: Drug: Nivolumab; Drug: Cisplatin; Drug: Hydroxyurea; Drug: 5-FU; Drug: Dexamethasone; Drug: Famotidine; Drug: Diphenhydramine; Drug: Paclitaxel; Radiation: Chemoradiotherapy

INTERVENTIONS:
Drug: nab-paclitaxel — All enrolled patients will receive three 21-day cycles of nab-paclitaxel (100 mg/m2 on days 1, 8, 15; 9 doses total)
  Other Names: nanoparticle albumin-bound paclitaxel; Abraxane
  Arms: Induction Chemotherapy
Drug: Carboplatin — All enrolled patients will receive three 21-day cycles of carboplatin (AUC 6 on day 1; 3 doses total).
  Other Names: paraplatin
  Arms: Induction Chemotherapy
Drug: Nivolumab — All enrolled patients will receive three 21-day cycles of nivolumab (360 mg on days 1; 3 doses total).
  Adjuvant nivolumab will be offered to all patients for 6-months post completion of locoregional therapy for a total of 7 doses.
  Other Names: Opdivo
Drug: Cisplatin — Cisplatin will be given on an every 3 weeks basis at a dose of 100 mg/m2 IV over 3-4 hrs day 1 (or 2) and 22 (or 23). Only for patients on the Intermediate Dose Arm and additionally on day 43 (or 44) for patients on the Regular Dose Arm.
  Other Names: platinol
  Arms: Intermediate De-escalation Arm (IDA); Regular Dose Arm (RDA)
Drug: Hydroxyurea — Patients on the Intermediate or Regular Dose Arms will receive chemoradiation for 3-5 cycles (6-10 weeks). On day 0 patients will start hydroxyurea at 500 mg PO q 12 hours x 6 days (11 doses). The first daily dose of hydroxyurea on days 1 - 5 is given 2 hours prior to the first fraction of daily radiotherapy.
  Arms: Intermediate De-escalation Arm (IDA); Regular Dose Arm (RDA)
Drug: 5-FU — Patients on the Intermediate or Regular Dose Arms will receive chemoradiation for 3-5 cycles (6-10 weeks). On day 0 at 1800 patients will start continuous infusion of 5-FU at 600 mg/m2/day x 5 days (120 hours).
  Other Names: Adrucil; Carac
  Arms: Intermediate De-escalation Arm (IDA); Regular Dose Arm (RDA)
Drug: Dexamethasone — Patients on the Intermediate or Regular Dose Arms will receive chemoradiation for 3-5 cycles (6-10 weeks). On days 1-5 patients will receive dexamethasone 20 mg PO (IV) in am Day 1, 1 hr prior to paclitaxel
  Arms: Intermediate De-escalation Arm (IDA); Regular Dose Arm (RDA)
Drug: Famotidine — Patients on the Intermediate or Regular Dose Arms will receive chemoradiation for 3-5 cycles (6-10 weeks). On days 1-5 patients will receive famotidine 20 mg PO (IV) in am Day 1, 1 hr prior to paclitaxel.
  Other Names: pepcid
  Arms: Intermediate De-escalation Arm (IDA); Regular Dose Arm (RDA)
Drug: Diphenhydramine — Patients on the Intermediate or Regular Dose Arms will receive chemoradiation for 3-5 cycles (6-10 weeks). On days 1-5 patients will receive diphenhydramine 50 mg PO (IV) in am Day 1, 30 mins prior to paclitaxel.
  Other Names: benadryl
  Arms: Intermediate De-escalation Arm (IDA); Regular Dose Arm (RDA)
Drug: Paclitaxel — Patients on the Intermediate or Regular Dose Arms will receive chemoradiation for 3-5 cycles (6-10 weeks). On days 1-5 patients will start paclitaxel 100 mg/m2 after first RT fraction on day 1 of each cycle. Paclitaxel should be administered in 250 ml 0.9% NaCl over 60 minutes.
  Other Names: taxol
  Arms: Intermediate De-escalation Arm (IDA); Regular Dose Arm (RDA)
Procedure: Transoral robotic surgery (TORS) — Patients with low risk and small volume tonsillar disease (T1-T2, non-bulky N2A-N2B with ≤2 non-lower neck lymph nodes measuring ≤5 cm in size) or base of tongue disease (T1-2 with lateralized primary ≤3 cm, non-bulky N2A-N2B with ≤2 non-lower neck lymph nodes measuring ≤5 cm in size) who have ≥50% reduction by RECIST following induction chemotherapy will undergo TORS and selective nodal dissection. Patients may refuse TORS treatment. Patients will receive RT or TORS.
  Other Names: TORS
  Arms: Single Modality De-escalation Arm (SDA)
Radiation: Adjuvant RT — Patients with low risk, who do not qualify for TORS (due to volume of disease or poor visualization/access) or refuse TORS, who have ≥50% reduction by RECIST following induction chemotherapy will be given de-intensified treatment with radiation alone to 50 Gy. Patients will receive RT or TORS.
  Other Names: RT
  Arms: Single Modality De-escalation Arm (SDA)
Radiation: Chemoradiotherapy — Patients who have low risk disease with <50% but ≥30% reduction, or patients who have high risk disease and ≥50% reduction of tumor by RECIST with induction chemotherapy will receive CRT to 50 Gy with concurrent bolus cisplatin (x2 doses) or TFHX to 45 Gy (3 cycles).
  Patients who have low risk disease and <30% reduction of tumor, patients who have high risk disease and <50% reduction of tumor by RECIST, or any patient who has progressive disease with induction chemotherapy will receive CRT to 70 Gy with concurrent bolus cisplatin (x3 doses) or TFHX to 75 Gy (5 cycles).
  Other Names: CRT
  Arms: Intermediate De-escalation Arm (IDA); Regular Dose Arm (RDA)

SUMMARY:
Carboplatin, nab-paclitaxel, and nivolumab combination will be administered for three cycles of three weeks duration each. TORS or RT/CRT will be performed after induction chemotherapy (i.e. day 64 of therapy). Patients with low risk and small volume tonsillar disease (T1-T2, non-bulky N2A-N2B with ≤2 non-lower neck lymph nodes measuring ≤5 cm in size) or base of tongue disease (T1-2 with lateralized primary ≤3 cm, non-bulky N2A-N2B with ≤2 non-lower neck lymph nodes measuring ≤5 cm in size) who have ≥50% reduction by RECIST following induction chemotherapy will undergo TORS and selective nodal dissection. De-intensified adjuvant RT will be given for adverse pathologic features. Patients may refuse TORS treatment.

Patients with low risk, who do not qualify for TORS (due to volume of disease or poor visualization/access) or refuse TORS, who have ≥50% reduction by RECIST following induction chemotherapy will be given de-intensified treatment with radiation alone to 50 Gy.

Before induction chemotherapy, patients will undergo examination under anesthesia and direct laryngoscopy to tattoo and photograph the primary tumor to plan the post-induction resection. Adjuvant nivolumab will be offered to all patients for 6-months post completion of definitive therapy (7 doses given as a flat dose of 480mg, every four weeks).

DETAILED DESCRIPTION:
A phase II trial in human papillomavirus (HPV)-positive oropharyngeal squamous cell cancer (as determined by p16 immunohistochemistry with confirmatory ISH or PCR) to determine radiologic response to induction chemotherapy with nivolumab. Patients will undergo evaluation by a multidisciplinary team prior to risk assessment. The patients will be assigned to high or low risk groups based on tumor size, lymph node involvement, and smoking history. Patients will be assigned to treatment with induction chemotherapy with carboplatin, nab-paclitaxel, and nivolumab. Radiologic response to induction chemotherapy according to RECIST measurement of tumor shrinkage will then be used for therapeutic stratification of locoregional therapy, consisting of either transoral robotic surgery (TORS) or radiation with or without chemotherapy. Patients with low risk disease (see table above) and small volume tonsillar/BOT disease (T1-2 primary, non-bulky N2A-N2B nodal status) who have ≥50% reduction by RECIST following induction chemotherapy will undergo TORS for primary site resection and selective nodal dissection as a definitive treatment if technically feasible with adjuvant radiation for adverse pathologic features. Patients with other low risk tumors e.g. with higher volume disease, or who refuse surgery, who also have ≥50% reduction by RECIST following induction chemotherapy will be given de-intensified treatment with radiation alone to 50 Gy (no chemotherapy). Patients with low risk features and <50% but ≥30% reduction OR high risk features (T4, bulky N2B or N2C-N3, >10 pack-years tobacco use) with ≥50% reduction will receive de-intensified chemoradiation with concurrent cisplatin-RT to 50 Gy (5 weeks) or TFHX to 45 Gy (3 cycles/6 weeks). Patients with low risk features and <30% reduction OR high risk disease with <50% reduction or any patients with progressive disease during induction chemotherapy will undergo chemoradiotherapy with concurrent cisplatin-RT to 70 Gy (7 weeks) or TFHX to 75 Gy (5 cycles/10 weeks). Patients with both high and low risk features who have ≥50% reduction will receive locoregional therapy targeting the pre-chemotherapy extent of disease only. Adjuvant nivolumab will be offered to all patients for 6-months post completion of definitive therapy (7 doses given as a flat dose of 480mg, every four weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed HPV-positive head and neck squamous cell carcinoma of the oropharynx. Confirmed HPV-positive disease of other subsites are uncommon but also eligible.
* HPV testing must be compliant with the following criteria:
* p16 IHC positivity is sufficient to enroll and initiate treatment (p16 IHC interpretation to follow guidelines by Jordan and Lingen et al89).
* p16 IHC positivity is to be validated using an HPV PCR during the induction phase. This is essential as HPV genotype influences treatment arm allocation, with non-HPV16 HPV strains being considered high risk.
* Availability of ≥10 unstained 5 micron slides (to be provided to HTRC at the University of Chicago). Patients who cannot fulfill this requirement will need to undergo a new biopsy prior to enrollment on study.
* Patients must be at least 18 years of age.
* Patients with AJCC (7th edition, 2010) N2-N3 nodal disease or T3-T4 primary tumor.
* Measurable disease (either primary site and/or nodal disease) by RECIST 1.1 criteria.
* No previous radiation or chemotherapy for a head and neck cancer.
* No complete surgical resection for a head and neck cancer within 8 weeks of enrollment (although lymph node biopsy including excision of an individual node with presence of residual nodal disease, or surgical biopsy/excision of the tumor with residual disease is acceptable).
* ECOG performance status 0-1 (Karnofsky greater than or equal to 80%).
* Normal Organ Function
* Leukocytes ≥3000/mm3,
* platelets ≥100,000/mm3,
* absolute neutrophil count ≥1,500,
* hemoglobin >9.0 gm/dL,
* AST and ALT <2.5 X ULN
* alkaline phosphatase <2.5 X ULN
* albumin >2.9 gm/dL, 29 Version Date: 12/28/2016
* total bilirubin ≤1.5 mg/dl,
* creatinine clearance >45 mL/min (or SCr <1.5 mg/dL), normal within 2 weeks prior to start of treatment.
* The standard Cockcroft and Gault formula or the measured glomerular filtration rate must be used to calculate CrCl for enrollment or dosing
* Patients must sign a study-specific informed consent form prior to study entry. Patients should have the ability to understand and the willingness to sign a written informed consent document.
* Age, Sex, and Reproductive Status:

  1. Men and women, ages > 18.
  2. Women of childbearing potential (WOCBP=premenopausal woman capable of becoming pregnant) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
  3. Women must not be breastfeeding.
  4. WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 5 half-lives of study drug(s) plus 30 days (duration of ovulatory cycle) for a total of 23 weeks post-treatment completion.
  5. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 5 half-lives of study drug(s) plus 90 days (duration of sperm turnover) for a total of 31 weeks post treatment completion.
  6. Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, they must still undergo pregnancy testing as described in this section.
* Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of <1% when used consistently and correctly.
* At a minimum subjects must agree to the use of one method of highly effective contraception as listed below:

HIGHLY EFFECTIVE METHODS OF CONTRACEPTION

* Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants and intrauterine devices (IUDs) such as Mirena® by WOCBP subject or male subject's WOCBP partner
* IUDs, such as ParaGard®
* Tubal ligation
* Vasectomy 30 Version Date: 12/28/2016
* Complete Abstinence*

  * *Complete abstinence is defined as complete avoidance of heterosexual intercourse and is an acceptable form of contraception for all study drugs. Female subjects must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence.

Subjects are encouraged to use two methods of contraception, with one method being highly effective and the other method being either highly effective or less effective as listed below:

LESS EFFECTIVE METHODS OF CONTRACEPTION

* Diaphragm with spermicide
* Cervical cap with spermicide
* Vaginal sponge
* Male condoms and spermicide
* Male condom without spermicide
* Progestin only pills by WOCBP subject or male subject's WOCBP partner
* Female condom*

  * *A male and female condom must not be used together

Exclusion Criteria:

* Unequivocal demonstration of distant metastases (M1 disease).
* Unidentifiable primary site.
* Intercurrent medical illnesses which would impair patient tolerance to therapy or limit survival. Including but not limited to ongoing or active infection, immunodeficiency, symptomatic congestive heart failure, pulmonary dysfunction, cardiomyopathy, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance.
* Pregnant and nursing women are excluded because of the potential teratogenic effects and potential unknown effects on nursing newborns (please see above paragraph under inclusion criteria regarding WOCBP) 31 Version Date: 12/28/2016
* Prior surgical therapy other than incisional/excisional biopsy or organ-sparing procedures such as debulking of airway-compromising tumors. Residual measurable tumor is required for enrollment on study as outlined above
* Patients receiving other investigational agents.
* Peripheral neuropathy >grade 1
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy in excess of physiologic dose or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active tuberculosis (Bacillus Tuberculosis infection)
* Has hypersensitivity to nivolumab or any other drug used in this protocol.
* Has had a prior systemic anti-cancer treatment within the last 8 weeks
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer or any tumors that are not likely to influence live expectancy in the subsequent 3 years without active treatment (e.g. low grade prostate cancer in absence of therapy).
* Has active autoimmune disease that has required systemic treatment in the past year (i.e. with use of steroids or immunosuppressive drugs). Replacement therapy e.g. levothyroxine, insulin, or physiologic corticosteroid doses for adrenal or pituitary insufficiency, etc. are not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has a history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected). However, if eradicated patient is eligible.
* Has received a live vaccine within 28 days of planned start of study therapy. o Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed within 28 days prior to initiation of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everett Vokes, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Rosenberg AJ, Agrawal N, Juloori A, Cursio J, Gooi Z, Blair E, Chin J, Ginat D, Pasternak-Wise O, Hasina R, Starus A, Jones FS, Izumchenko E, MacCracken E, Wolk R, Cipriani N, Lingen MW, Pearson AT, Seiwert TY, Haraf DJ, Vokes EE. Neoadjuvant Nivolumab Plus Chemotherapy Followed By Response-Adaptive Therapy for HPV+ Oropharyngeal Cancer: OPTIMA II Phase 2 Open-Label Nonrandomized Controlled Trial. JAMA Oncol. 2024 Jul 1;10(7):923-931. doi: 10.1001/jamaoncol.2024.1530. PMID 38842838

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Modality De-escalation Arm (SDA): Patients with low risk, who do not qualify for TORS (due to volume of disease or poor visualization/access) or refuse TORS, who have ≥50% reduction by RECIST following induction chemotherapy will be given de-intensified treatment with radiation alone to 50 G.
  Nivolumab: All enrolled patients will receive three 21-day cycles of nivolumab (360 mg on days 1; 3 doses total).
  Adjuvant nivolumab will be offered to all patients for 6-months post completion of locoregional therapy for a total of 7 doses.
  Transoral robotic surgery (TORS): Patients with low risk and small volume tonsillar disease (T1-T2, non-bulky N2A-N2B with ≤2 non-lower neck lymph nodes measuring ≤5 cm in size) or base of tongue disease (T1-2 with lateralized primary ≤3 cm, non-bulky N2A-N2B with ≤2 non-lower neck lymph nodes measuring ≤5 cm in size) who have ≥50% reduction by RECIST following induction chemotherapy will undergo TORS and selective nodal dissection. Patients may refuse TORS treatment. Patients will receive RT or TORS.
  Adjuvant RT: Patients with low risk, who do not qualify for TORS (due to volume of disease or poor visualization/access) or refuse TORS, who have ≥50% reduction by RECIST following induction chemotherapy will be given de-intensified treatment with radiation alone to 50 Gy. Patients will receive RT or TORS.
- Intermediate De-escalation Arm (IDA): Patients who have high risk disease and ≥50% reduction of tumor by RECIST with induction chemotherapy will receive CRT to 50 Gy with concurrent bolus cisplatin (x2 doses) or TFHX to 45 Gy (3 cycles).
Period: Overall Study
Arm/Group | Single Modality De-escalation Arm (SDA) | Intermediate De-escalation Arm (IDA) | Regular Dose Arm (RDA)
Started | 28 | 34 | 10
Completed | 28 | 34 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Modality De-escalation Arm (SDA): Radiation alone or transoral robotic surgery.
- Intermediate De-escalation Arm (IDA): TFHX (paclitaxel (100mg/m2 on day 1), 5-fluorouracil continuous infusion (600mg/m2/d on days 0-5), and hydroxyurea (500mg orally twice daily on days 0-5 with 11 doses per cycle )or cisplatin.
- Regular Dose Arm (RDA): Regular dose chemoradiotherapy and TFHX (paclitaxel (100mg/m2 on day 1), 5-fluorouracil continuous infusion (600mg/m2/d on days 0-5), and hydroxyurea (500mg orally twice daily on days 0-5 with 11 doses per cycle )or cisplatin.
- Total: Total of all reporting groups
Arm/Group | Single Modality De-escalation Arm (SDA) | Intermediate De-escalation Arm (IDA) | Regular Dose Arm (RDA) | Total
Number analyzed (Participants) | 28 | 34 | 10 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (8.5) | 64.4 (10.4) | 59.6 (7.9) | 61.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 0 | 6
  Male | 25 | 31 | 10 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 28 | 32 | 9 | 69
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 4
  White | 26 | 29 | 8 | 63
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 28 | 34 | 10 | 72

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Tumor Shrinkage (%) to Measure the Deep Response Rate (DRR)
Description: DRR is defined as ≥50% tumor shrinkage by RECIST 1.1. We will evaluate the overall percentage of patients treated with dose-reduced radiotherapy or TORS to determine the tumor shrinkage based on treatment received.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Single Modality De-escalation Arm (SDA): Radiotherapy alone or transoral robotic surgery
- Intermediate De-escalation Arm (IDA): TFHX (paclitaxel (100mg/m2 on day 1), 5-fluorouracil continuous infusion (600mg/m2/d on days 0-5), and hydroxyurea (500mg orally twice daily on days 0-5 with 11 doses per cycle) or Cisplatin
- Regular Dose Arm (RDA): Regular dose chemoradiotherapy and TFHX (paclitaxel (100mg/m2 on day
  1), 5-fluorouracil continuous infusion (600mg/m2/d on days 0-5), and hydroxyurea (500mg orally twice daily on days 0-5 with 11 doses per cycle) or Cisplatin
Arm/Group | Single Modality De-escalation Arm (SDA) | Intermediate De-escalation Arm (IDA) | Regular Dose Arm (RDA)
Number analyzed (Participants) | 28 | 34 | 10
Participants | 25 | 26 | 0

2. Secondary Outcome: Number of Patients With Adverse Events
Description: All recorded adverse events will be listed and tabulated by system organ class, preferred term and treatment. Vital signs and clinical laboratory test results will be listed and summarized by treatment. Any significant physical examination findings, and clinical laboratory results will be listed. ECG readings will be evaluated by the investigator and abnormalities, if present, will be listed.
Time Frame: 24 months
Population: Counts below represent the number of patients in each treatment group with any adverse event. More detailed information is provided in the adverse events section.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Modality De-escalation Arm (SDA) | Intermediate De-escalation Arm (IDA) | Regular Dose Arm (RDA)
Number analyzed (Participants) | 28 | 34 | 10
Participants | 27 | 29 | 10

3. Secondary Outcome: 2 Year Progression-free Survival (PFS)
Description: The percent of patients who are alive and did not progress after two years.
Time Frame: From start date of therapy to the date of first documented disease progression or death from any cause, whichever may come first, assessed up to 24 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Single Modality De-escalation Arm (SDA) | Intermediate De-escalation Arm (IDA) | Regular Dose Arm (RDA)
Number analyzed (Participants) | 28 | 34 | 10
percentage of patients | 99 [77 to 99] | 88 [71 to 95] | 100 [100 to 100]

4. Secondary Outcome: 2 Year Overall Survival (OS)
Description: The percent of patients that are alive after 2 years of follow up. Rates are estimated using Kaplan-Meier survival methods.
Time Frame: From start date of therapy to the date of documented death, assessed up to 24 months
Measure: Number (95% Confidence Interval); unit: percentage of patients in each arm
Arm/Group | Single Modality De-escalation Arm (SDA) | Intermediate De-escalation Arm (IDA) | Regular Dose Arm (RDA)
Number analyzed (Participants) | 28 | 34 | 10
percentage of patients in each arm | 96 [77 to 99] | 91 [74 to 97] | 87 [39 to 98]

5. Secondary Outcome: 2 Year Rates of Locoregional Control
Description: Time to locoregional failure rates will be estimated by the Kaplan-Meier methodology and comparisons will be made using the log-rank test.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Single Modality De-escalation Arm (SDA) | Intermediate De-escalation Arm (IDA) | Regular Dose Arm (RDA)
Number analyzed (Participants) | 28 | 34 | 10
percentage of patients | 96 [77 to 99] | 96 [79 to 99] | 100 [100 to 100]

6. Secondary Outcome: 2 Year Rates of Distant Control
Description: Time to distant failure rates will be estimated by the Kaplan-Meier methodology and comparisons will be made using the log-rank test.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Single Modality De-escalation Arm (SDA) | Intermediate De-escalation Arm (IDA) | Regular Dose Arm (RDA)
Number analyzed (Participants) | 28 | 34 | 10
percent of participants | 100 [100 to 100] | 97 [80 to 99] | 100 [100 to 100]

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Single Modality De-escalation Arm (SDA) | Intermediate De-escalation Arm (IDA) | Regular Dose Arm (RDA)
All-Cause Mortality (participants affected / at risk) | 1/28 | 3/34 | 1/10
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/34 | 0/10
Other Adverse Events (participants affected / at risk) | 27/28 | 29/34 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Modality De-escalation Arm (SDA) (N=28) | Intermediate De-escalation Arm (IDA) (N=34) | Regular Dose Arm (RDA) (N=10)
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 11 (11) | 13 (17) | 1 (3) — Anemia
Blood and lymphatic system disorders- other (Blood and lymphatic system disorders) | 5 (7) | 2 (2) | 1 (1)
Febrile neutropena (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Atrial Afribilation (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Chest pain- cardiac (Cardiac disorders) | 1 (2) | 1 (2) | 0 (0)
Heart Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 3 (4) | 0 (0)
Cardiac disorders other (Cardiac disorders) | 3 (3) | 3 (4) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 8 (9) | 6 (6) | 1 (1)
Hearing impared (Ear and labyrinth disorders) | 4 (4) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 5 (5) | 2 (2) | 3 (4)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (3) | 2 (2) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders other (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 18 (23) | 19 (22) | 8 (9)
Diarrhea (Gastrointestinal disorders) | 9 (10) | 14 (21) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 12 (13) | 6 (6) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 10 (15) | 18 (21) | 4 (4)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 13 (36) | 19 (64) | 5 (18)
Nausea (Gastrointestinal disorders) | 23 (37) | 21 (34) | 6 (9)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 7 (11) | 14 (23) | 6 (8)
Rectal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Salivary duct inflammation (Gastrointestinal disorders) | 4 (7) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 9 (13) | 6 (7) | 4 (5)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 9 (15) | 3 (3) | 2 (3)
Chills (General disorders) | 3 (3) | 2 (2) | 0 (0)
Edema face (General disorders) | 2 (2) | 1 (1) | 1 (2)
Edema limbs (General disorders) | 3 (3) | 3 (4) | 2 (2)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 24 (51) | 25 (51) | 8 (15)
Fever (General disorders) | 7 (7) | 3 (5) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 2 (2) | 0 (0)
Gait disturbance (General disorders) | 2 (2) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Localized edema (General disorders) | 3 (3) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0) | 0 (0)
Neck edema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 4 (5) | 2 (2) | 4 (7)
General disorders and administration site conditions - Other (General disorders) | 3 (3) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Immune system disorders - Other (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 2 (3) | 0 (0) | 1 (1)
Small intestine infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Stoma site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 11 (13) | 17 (35) | 5 (11)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (5) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 10 (15) | 4 (8) | 1 (1)
Alkaline phosphatase increased (Investigations) | 7 (7) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (9) | 1 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 3 (4) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (5) | 4 (5) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 5 (5) | 1 (1)
Weight gain (Investigations) | 1 (1) | 1 (1) | 0 (0)
Weight loss (Investigations) | 4 (8) | 3 (6) | 2 (2)
White blood cell decreased (Investigations) | 10 (12) | 7 (8) | 4 (4)
Investigations - Other (Investigations) | 0 (0) | 2 (2) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 11 (13) | 13 (23) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4) | 4 (5) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 2 (2)
Trismus (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 7 (8) | 5 (8) | 3 (6)
Dysarthia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 17 (28) | 13 (14) | 2 (3)
Headache (Nervous system disorders) | 7 (8) | 6 (6) | 2 (4)
Paresthesia (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 5 (13) | 6 (11) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (10) | 10 (13) | 6 (10)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
Anxiety (Eye disorders) | 2 (2) | 3 (4) | 1 (2)
Confusion (Psychiatric disorders) | 1 (3) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 7 (8) | 7 (8) | 2 (3)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (4) | 3 (3) | 2 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1) | 3 (4) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 6 (10) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (5) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (5) | 2 (2)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (5) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 3 (5)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 8 (9) | 4 (4)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (7) | 5 (7) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (5) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (9) | 4 (5) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 7 (11) | 4 (6) | 1 (1)
Hypertension (Vascular disorders) | 5 (12) | 5 (5) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 5 (5) | 2 (3)
Lymphedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT03107182/Prot_SAP_000.pdf